CLINICAL TRIAL: NCT06674252
Title: A Randomized Controlled Multicenter Study on the Improvement of Postoperative Symptoms and Survival Benefits of Modified Bufei Decoction in Elderly Patients With Lung Cancer Undergoing Radical Surgery
Brief Title: A Study on the Improvement of Postoperative Symptoms and Survival Benefits of Modified Bufei Decoction in Elderly Patients With Lung Cancer Undergoing Radical Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JWBF-1
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancers
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jiawei Bufei Tang (Experimental): Oral administration of Jiawei Bufei Tang granules for 28 days, twice a day, 1 packet each time, and the medication must be taken with water.
  Interventions: Other: Jiawei Bufei Tang granules
- Placebo granules (Placebo Comparator): Take placebo granules orally for 28 days, twice a day, 1 pack each time, and the medication must be taken with water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Other: Jiawei Bufei Tang granules — Jiawei Bufei Tang is a traditional Chinese medicine formula applied by Professor Li Pingping to patients with lung cancer and qi yin deficiency syndrome. It consists of Huangqi, Codonopsis pilosula, Schisandra chinensis, Rehmannia glutinosa, Ziyuan, Mulberry bark, Snake berry, Half branch Lotus, White Hedyotis diffusa, etc. Bu Fei Tang is derived from the Yuan Dynasty's "Yong Lei Ling Fang" and consists of six ingredients: ginseng, astragalus, schisandra, Radix Rehmanniae, Ziyuan, and mulberry bark. It is mainly used to treat cough caused by lung qi deficiency. Jiawei Bufei Tang adds white Hedyotis diffusa, Scutellaria barbata, and snake berry to the original formula. White Hedyotis diffusa is more effective in dispelling carbuncles and detoxifying, Scutellaria barbata is more effective in dispelling phlegm and diuresis, and snake berry is more effective in dispelling scrofula and dispersing nodules, increasing the effect of clearing heat and detoxifying. This formula is particularly e
  Arms: Jiawei Bufei Tang
Drug: Placebo — placebo
  Arms: Placebo granules

SUMMARY:
This is a randomized double-blind placebo-controlled phase II clinical study that included patients with symptoms such as cough, shortness of breath, and fatigue after lung cancer resection surgery. They were given orally modified Bufei Tang granules twice a day for 28 days, with one packet taken orally with water. Using the MDASI-TCM symptom scoring system, evaluate the scores of symptoms such as cough, shortness of breath, and fatigue before and after the experiment, and calculate the difference in scores between the control group and the experimental group before and after the experiment.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial to verify the effectiveness of the traditional Chinese medicine compound Jiawei Bufei Tang in improving postoperative clinical symptoms in elderly lung cancer patients and providing effective treatment methods for improving patients' quality of life.

1. Research Design: A multicenter, randomized double-blind placebo-controlled study was conducted, in which eligible subjects were randomly assigned to a treatment group and a control group in a 1:1 ratio, with 87 cases in each group.
2. The process of participant participation in the experiment The composition of Jiawei Bu Fei Tang includes Huangqi, Codonopsis pilosula, Schisandra chinensis, Rehmannia glutinosa, Ziyuan, Mulberry bark, Snake berry, Half branch lotus, White Hedyotis diffusa, Bai Qian, and Platycodon grandiflorum. A traditional Chinese medicine placebo is formulated with caramel color, dextrin, and bittering agent to create a placebo with an appearance and taste similar to the treatment group's medication. Both the therapeutic drug and placebo were tested using independently packaged non decoction granules produced by the same company and batch.

On the 7th day after surgery, patients were screened and evaluated using the MDASI-TCM scale. Subjects with postoperative symptoms such as fatigue, cough, and shortness of breath who met the inclusion criteria but did not meet the exclusion criteria were included in the clinical study and randomly assigned to receive oral medication treatment in a 1:1 ratio.

On the day of inclusion, the patient was randomized and successfully received the trial medication, with the first oral administration of traditional Chinese medicine within 24 hours.

Treatment group (Modified Bufei Decoction):

Usage of traditional Chinese medicine: Take orally 1 bag/time of Jiawei Bufei Tang, twice a day, starting from the 7th day after surgery (the day of enrollment), for 28 consecutive days.

Control group (placebo):

Usage of placebo: Take 1 bag of placebo orally, twice a day, starting from the 7th day after surgery (the day of enrollment), for 28 consecutive days.

If the subject experiences discomfort during the medication process, unblinding or withdrawal from the study can be based on the researcher's judgment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with postoperative lung cancer who have clear histological or cytological diagnosis.

  * Age ≥ 65 years old, both male and female are eligible. According to the MDASI-TCM scale evaluation, any of the three symptoms of cough, fatigue, and shortness of breath should score ≥ 4 points, or the sum of the three should score ≥ 6 points.

    * The heart function is basically normal; ALT/AST is within 2 times the normal value; SCr is within the normal range.

Traditional Chinese medicine syndrome differentiation is characterized by deficiency of both lungs and kidneys.

Exclusion Criteria:

* Patients with severe pulmonary infections. ⑵. Patients with mental illness. ⑶. Patients with depression.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
MDASI-TCM scale | 28 days
  The symptom score results of the MDASI-TCM scale between the oral Chinese medicine group and the placebo group after 28 days of medication.

SECONDARY OUTCOMES:
QLQ-C30 scale | 28 days
  Compare the QLQ-C30 scale scores before and after the trial between the modified Bufei Decoction group and the placebo group
CGA assessment | 28 days
  Compare the CGA assessment results of elderly patients before and after the trial between the modified Bufei Decoction group and the placebo group
DFS | 28 days
  Record the difference in DFS between the modified Bufei Decoction group and the placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing cancer hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes